CLINICAL TRIAL: NCT07232121
Title: A Phase 1 Double-Blind, Randomized, Placebo-Controlled, Single Ascending Dose Study to Evaluate Safety, Tolerability, Pharmacokinetics, Immunogenicity and Pharmacodynamics of DF5112 in Healthy Adult Participants
Brief Title: A Study to Evaluate the Safety of Increasing Doses of DF5112 in Healthy Adults
Acronym: DF5112
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dragonfly Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: DF5112-001
Record Dates: First submitted 2025-11-13; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants; Healthy Adult Females; Healthy Adult Male; Healthy; Volunteer
Keywords: Healthy Volunteer; Healthy Participant

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DF5112 (Experimental): Single dose of DF5112 administered either via IV or SC
  Interventions: Drug: DF5112
- Placebo (Placebo Comparator): Single dose of placebo administered either via IV or SC
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DF5112 — DF5112 administered IV or SC
  Arms: DF5112
Other: Placebo — Placebo administered IV or SC.
  Arms: Placebo

SUMMARY:
This is a double-blind, randomized, placebo-controlled, single ascending dose (SAD) study to evaluate safety, tolerability, pharmacokinetics (PK), immunogenicity and pharmacodynamics (PD) of DF5112 in healthy adult participants. A total of 64 participants are planned to be randomized into 8 cohorts. Additional cohorts at intermediate dose levels may be evaluated. Each cohort will include 8 healthy participants randomized to receive DF5112 or placebo through intravenous (IV) or subcutaneous (SC) administration. Following dose administration participants will be confined at the clinical research unit for observation for approximately 1 week and then will return for subsequent pre-identified follow up visits through at least Day 29, Day 57, or Day 85 (length of follow-up is determined by the cohort).

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female participants aged 18 to 55 years (inclusive) at the time of informed consent.
* Body mass index (BMI) between ≥ 18.0 and ≤ 32.0 kg/m2 and body weight ≥ 45 kg.
* At the discretion of the Principal Investigator (PI) or designee, in good general health, with no significant medical history, and have no clinically significant abnormalities on physical examination at Screening and/or before the first administration of IP.
* Clinical laboratory values within normal range as specified by the testing laboratory, unless deemed not clinically significant by the PI or designee.

Key Exclusion Criteria:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrinological, hematological, or neurological disorders that, in the opinion of the PI or designee, are capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention; or interfering with the interpretation of data.
* History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system treated or untreated within the past 5 years, regardless of whether there is evidence of local recurrence or metastases (except for squamous and basal cell carcinoma of the skin or actinic keratoses that have been treated with no evidence of recurrence in the past 12 weeks; carcinoma in situ of the cervix or non-invasive malignant colon polyps that have been removed).
* History of or evidence of recurrent or chronic bacterial or fungal infections including those of the skin, vagina, oral cavity, etc., or systemic fungal infection.
* History of unexplained, recurrent infection, or infection requiring treatment with systemic antibiotics within 90 days prior to dosing on Day 1.
* Active oral infection.
* Acute illness (e.g. common cold) within 2 weeks prior to Screening, or seasonal influenza or COVID within 4 weeks prior to Screening.
* History of latent or active tuberculosis that has not been adequately treated, at the discretion of the PI or designee.
* Positive or inconclusive hepatitis B or hepatitis C based antibody tests at Screening.
* Positive human immunodeficiency virus (HIV) antibody test at Screening.
* History of severe allergy, hypersensitivity reaction, or anaphylaxis to drugs or human proteins or components of the study drug formulation used in this study.
* Any vaccination within 1 month of Day 1 and planned within 1 month post Day 1. Any live or attenuated vaccine within 1 month prior to Day 1 and planned within 3 months post Day 1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | From Day 1 dosing to end of study at Day 29, 57, or 85 (depending on cohort)

SECONDARY OUTCOMES:
To evaluate the PK of single ascending doses of DF5112 administered by IV or SC injection | From Day 1 dosing to end of study at Day 29, 57, or 85 (depending on cohort)
  PK parameter: Area Under the Concentration Curve (AUC)
Incidence and titer of Anti-Drug Antibodies | From Day 1 dosing to end of study at Day 29, 57, or 85 (depending on cohort)

CONTACTS AND LOCATIONS:
Locations (1):
- Scientia Clinical Research Ltd, Sydney, New South Wales, Australia